CLINICAL TRIAL: NCT04919161
Title: Unblinded Quasi-Randomized Pilot Study Exploring the Benefits of the ZeroG TRiP System to Improve Patient Balance Following an Acute Stroke
Brief Title: Explorations of the Benefits of the ZeroG TRiP System to Improve Balance in Patients Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaylord Hospital, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201901Ber
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Balance; Distorted
Keywords: Stroke Rehabilitation; Postural Balance; Gait and Ambulation; Balance Perturbation; Postural Perturbation; Body Weight Support System; Occupational Therapy; Physical Therapy; Long Term Acute Care Hospital; Berg Balance Scale; Activities Specific Balance Confidence Scale; Balance Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Quasi-randomized controlled pilot study evaluating the efficacy of a recently developed, not yet reported, balance perturbation module for the ZeroG body weight support system known Training Responses in Postural rehabilitation (TRiP).
Masking Description: Participants and care providers are unable to be masked to the intervention arm due to the nature of the study. As data was extracted, investigators were unable to blind the data prior to exporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Body weight support system control group (Active Comparator): In this arm, participants will undergo their normal physical therapy treatment while using the ZeroG body weight support system.
  Interventions: Device: Body weight support system control group
- Body weight support system with balance perturbations (Experimental): Similar to the control group arm, participants will undergo their normal physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions.
  Interventions: Device: Body weight support system with balance perturbations
- Historical Standard of Care control (No Intervention): Retrospective anonymized Berg Balance Score data of stroke inpatients was collected from an institutional report for fiscal year 2018. 2018 was chosen as it preceded the implementation of the ZeroG body weight support system and reflects a no-intervention control baseline. This data was then filtered to show only patients with a Berg score of 21 or greater to match the study's inclusion criteria.

INTERVENTIONS:
Device: Body weight support system control group — The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
  Other Names: ZeroG; BWSS; BWSS control
  Arms: Body weight support system control group
Device: Body weight support system with balance perturbations — The BWSS with balance perturbations group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.In addition, this arm will receive eight balance perturbations, two in each direction (lateral, anterior, and posterior) each session. BWSS-P participants will start at perturbation level "one" and progress up to level "ten" as appropriate. Each session, the perturbation level will be set based on the participant's progress.
  Other Names: ZeroG with training response in postural rehabilitation; BWSS-P; BWSS+P
  Arms: Body weight support system with balance perturbations

SUMMARY:
Strokes are neurological events that can lead to devastating physical and cognitive deficits, such as the inability to ambulate, impaired balance regulation, and loss of coordination. Due to the physical and cognitive deficits experienced following a stroke, many require admission to an inpatient rehabilitation facility to maximize their independence before returning to the home setting. The ability to walk, stand, climb stairs, and other mobility-related functional tasks, are critical components of achieving this functional independence. However, it is often difficult for post-stroke patients with balance impairments to safely practice balance and gait training without putting both therapists and patients at risk for injury. Incorporating robotic technologies to neurological rehabilitation can play a critical role in delivering safe and effective gait and balance therapy.

Body-weight support systems (BWSSs) unload paretic lower limbs, patients with gait impairments can practice a higher repetition of steps in a safe, controlled manner. As participants perform gait training, these systems support the participant's body-weight, permitting those with excessive weakness and poor coordination, to ambulate and perform more intensive therapy sessions sooner in their recovery, with minimal risk injurious fall. In addition to BWSSs, balance perturbation systems, which purposefully unbalance participants so to rehabilitate their postural control, have been used to improve gait and balance-control after stroke, or other age and disease related balance impairments.

The goal of this study was to evaluate the efficacy of a recently developed, not yet reported, balance perturbation module for the ZeroG BWSS. This new balance perturbation training module is directly integrated into the ZeroG BWSS and allows for the direct induction of safe lateral, anterior, and/or posterior perturbations via a Wi-Fi-enabled handheld device. During both stationary and ambulatory activities, this system was used unbalance participants in order to train their balance-control and balance-reactions. The purpose of this pilot study was to determine if this newly developed BWSS balance perturbation system more effectively rehabilitates participant gait and balance after stroke than the standard BWSS protocol without perturbations.

DETAILED DESCRIPTION:
Body-Weight Support System Equipment and Interventions:

For this study, the BWSS used was the FDA listed ZeroG Gait and Balance System (Aretech, LLC, Ashburn, VA). ZeroG was first introduced to the investigators institution in September 2019. Unlike some BWSSs, this device is mounted on an overhead track that follows users during ambulation. Like other BWSSs, this system is designed to unload the users of up-to 200 pounds of their body weight while simultaneously protecting patients from falling. For this study, 10 pounds of participants' body-weight, the system minimum required to engage the BWSS, was continuously displaced. If a participant were to fall, the system would detect the change, decelerate, and stop the descent after a set distance; the fall distance was set between 8 to 12 inches for the purpose of this study. Unlike other BWSSs, a newly developed balance perturbation module known as the Training Responses in Postural rehabilitation or TRiP, is directly integrated to the ZeroG BWSS. This perturbation module is different than other systems as the balance perturbations are elicited directly through the BWSS and do not require a treadmill, tilt-table/shaking platform, or manual exertion by a. Further, they can be induced during normal gait and balance exercises during therapy. The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions. The BWSS with perturbation (BWSS-P) intervention group performed the same activities as the control group, with the addition of lateral, anterior, and posterior perturbations. Assistive devices and equipment were used during intervention sessions as recommended by the participant's primary therapist, including: canes, rolling walkers, hemi-walkers, and ankle-foot-orthoses (AFO), ankle support braces, and upper extremity slings.

Investigators administered perturbations using a Wi-Fi-enabled handheld device linked to the BWSS and these consisted of a sudden and brief assistive or resistive force in the desired direction. Lateral perturbations were issued while participants were in a static stance, while anterior and posterior perturbations were issued during ambulation; eight perturbations, two in each direction, were completed each session. All participants started at perturbation level "one" and progressed up to a maximum perturbation level of "ten" through the course of the study. The amount of force exerted at each perturbation level is pre-set by the manufacturer. The perturbation level (i.e. intensity or force) used each session was based on the participant's progress and observational analysis made by the investigator of the participants' response to the perturbation level. If the participant was able to tolerate the initial perturbation level without exhibiting a balance reaction, the perturbation level was incrementally increased until an appropriate balance reaction was exhibited. If a participant was unable to recover and elicited a fall response in the system, the perturbation level was decreased by one level to ensure patient safety, and the exercise repeated to reinforce the exercise mechanics and participant confidence.

Participants in both study groups received a total of eight treatment sessions over two weeks. As necessary, participants received up to two sessions in one day to ensure they completed the required eight sessions before discharge. These sessions were incorporated into the participants' regular care. Treatment sessions were broken into 30 minute blocks as it standard at the host facility. This time includes participant transportation, equipment set-up, and in the case of this study, donning the BWSS harness. On average, participants received 20 minutes of active time in the BWSS for each 30 minute treatment block. All sessions were analyzed equally despite the length of time in the BWSS.

Missing data:

When outcome measurements are missing due to early participant withdrawal, if the participant completed 50% or less of the study sessions, that participant's data was removed. If the participant completed greater than 50%, then that participant's data was analyzed as normal.

Data Analysis:

Data was analyzed using GraphPad Prism version 9.0.0 (GraphPad Software, San Diego, CA). To compare the observed proportion of males and females in the BWSS groups, a Binomial Test and Fisher's exact test were used. The 95% confidence intervals reported the proportion of males and females in the BWSS-P group were calculated using the Wilson-Brown Method. Berg Balance Scale (BBS) and Activities specific Balance Confidence measurement changes between the pre- and post-intervention were compared directly, as well as between groups. The degree of change made by each individual was shown by calculating the percent change: [((Post assessment) - (Pre assessment)) / (Pre assessment)] ×100% .

BBS data of stroke rehabilitation patients from fiscal year 2018 served as a historical standard of care (SOC) baseline control. The SOC data was sorted to consist of patients with initial BBS scores of 21 or greater and who were admitted and discharged before the launch of the institution's BWSS in September 2018. This resulted in the inclusion of retrospective BBS data from 30 patients. Shapiro-Wilk testing was first used to test for normality; if one or more of the data-sets in the group failed (p<0.05), nonparametric tests were used going forward. For hypothesis testing between two groups, unpaired or paired two-tailed Student's t-test were conducted as appropriate. When indicated by an F-test for variance (p<0.05), Welch's correction was applied for unequal standard deviations between groups. When comparing three or more groups, if one or more groups were abnormally distributed, non-parametric Kruskal-Wallis analysis of variation (ANOVA) test and Dunn's multiple comparison test for statistical hypothesis testing were used. When normally distributed, an Ordinary one-way ANOVA with a Tukey's multiple comparisons test for statistical hypothesis testing was used. If Brown-Forsythe's test for variance indicated the variance of the groups were significantly different (p<0.05), a Brown-Forsythe correction was applied and Dunnett's T3 multiple comparisons test for statistical hypothesis testing was used instead.

ELIGIBILITY:
Inclusion Criteria:

* Admission Berg Balance Scale score of 21 or greater
* 18 years of age or older
* Be able to understand and respond to simple verbal instructions in any language
* Be able to physically tolerate and actively participate in at least three, 30 minute weekly sessions in the ZeroG body weight support system

Exclusion Criteria:

* Cognitive deficits that would disrupt the ability to provide informed consent
* Admission Berg Balance Scale score less than 21
* Uncontrolled hypotension
* Uncontrolled hypertension
* Unstable skin structure (i.e. skin grafts, chest tubes)
* Unstable rib or lower extremity fractures
* Osteoporosis
* Active enteric infection control precautions
* New limb amputations
* Need for greater than 50% high flow oxygen
* Body weight greater than 450 pounds (structural limitations of the ZeroG body weight support system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Meyer, MS OTR/L, Principal Investigator — Gaylord Hospital
Locations (1):
- Gaylord Hospital, Wallingford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Copies of the study protocol will be provided upon request. Requests for copies of deidentified study data will considered on a case by case basis

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Alguren B, Lundgren-Nilsson A, Sunnerhagen KS. Functioning of stroke survivors--A validation of the ICF core set for stroke in Sweden. Disabil Rehabil. 2010;32(7):551-9. doi: 10.3109/09638280903186335. PMID 20136473
- [Background] Chen N, Xiao X, Hu H, Chen Y, Song R, Li L. Identify the Alteration of Balance Control and Risk of Falling in Stroke Survivors During Obstacle Crossing Based on Kinematic Analysis. Front Neurol. 2019 Jul 30;10:813. doi: 10.3389/fneur.2019.00813. eCollection 2019. PMID 31417488
- [Background] Forster A, Young J. Incidence and consequences of falls due to stroke: a systematic inquiry. BMJ. 1995 Jul 8;311(6997):83-6. doi: 10.1136/bmj.311.6997.83. PMID 7613406
- [Background] Legters K. Fear of falling. Phys Ther. 2002 Mar;82(3):264-72. No abstract available. PMID 11869155
- [Background] Landers MR, Oscar S, Sasaoka J, Vaughn K. Balance Confidence and Fear of Falling Avoidance Behavior Are Most Predictive of Falling in Older Adults: Prospective Analysis. Phys Ther. 2016 Apr;96(4):433-42. doi: 10.2522/ptj.20150184. Epub 2015 Aug 20. PMID 26294679
- [Background] Hidler J, Hamm LF, Lichy A, Groah SL. Automating activity-based interventions: the role of robotics. J Rehabil Res Dev. 2008;45(2):337-44. doi: 10.1682/jrrd.2007.01.0020. PMID 18566951
- [Background] Hidler J, Lum PS. The road ahead for rehabilitation robotics. J Rehabil Res Dev. 2011;48(4):vii-x. doi: 10.1682/jrrd.2011.02.0014. No abstract available. PMID 21674383
- [Background] Chien JE, Hsu WL. Effects of Dynamic Perturbation-Based Training on Balance Control of Community-Dwelling Older Adults. Sci Rep. 2018 Nov 22;8(1):17231. doi: 10.1038/s41598-018-35644-5. PMID 30467355
- [Background] Shimada H, Obuchi S, Furuna T, Suzuki T. New intervention program for preventing falls among frail elderly people: the effects of perturbed walking exercise using a bilateral separated treadmill. Am J Phys Med Rehabil. 2004 Jul;83(7):493-9. doi: 10.1097/01.phm.0000130025.54168.91. PMID 15213472
- [Background] Esmaeili V, Juneau A, Dyer JO, Lamontagne A, Kairy D, Bouyer L, Duclos C. Intense and unpredictable perturbations during gait training improve dynamic balance abilities in chronic hemiparetic individuals: a randomized controlled pilot trial. J Neuroeng Rehabil. 2020 Jun 17;17(1):79. doi: 10.1186/s12984-020-00707-0. PMID 32552850
- [Background] Steib S, Klamroth S, Gassner H, Pasluosta C, Eskofier B, Winkler J, Klucken J, Pfeifer K. Perturbation During Treadmill Training Improves Dynamic Balance and Gait in Parkinson's Disease: A Single-Blind Randomized Controlled Pilot Trial. Neurorehabil Neural Repair. 2017 Aug;31(8):758-768. doi: 10.1177/1545968317721976. Epub 2017 Jul 31. PMID 28758519
- [Background] Schinkel-Ivy A, Huntley AH, Aqui A, Mansfield A. Does Perturbation-Based Balance Training Improve Control of Reactive Stepping in Individuals with Chronic Stroke? J Stroke Cerebrovasc Dis. 2019 Apr;28(4):935-943. doi: 10.1016/j.jstrokecerebrovasdis.2018.12.011. Epub 2019 Jan 7. PMID 30630753
- [Background] Mansfield A, Aqui A, Danells CJ, Knorr S, Centen A, DePaul VG, Schinkel-Ivy A, Brooks D, Inness EL, Mochizuki G. Does perturbation-based balance training prevent falls among individuals with chronic stroke? A randomised controlled trial. BMJ Open. 2018 Aug 17;8(8):e021510. doi: 10.1136/bmjopen-2018-021510. PMID 30121600
- [Background] Hidler J, Brennan D, Black I, Nichols D, Brady K, Nef T. ZeroG: overground gait and balance training system. J Rehabil Res Dev. 2011;48(4):287-98. doi: 10.1682/jrrd.2010.05.0098. PMID 21674384
- [Background] Anggelis E, Powell ES, Westgate PM, Glueck AC, Sawaki L. Impact of motor therapy with dynamic body-weight support on Functional Independence Measures in traumatic brain injury: An exploratory study. NeuroRehabilitation. 2019 Dec 18;45(4):519-524. doi: 10.3233/NRE-192898. PMID 31868690
- [Background] Hutchinson LA, De Asha AR, Rainbow MJ, Dickinson AWL, Deluzio KJ. A comparison of centre of pressure behaviour and ground reaction force magnitudes when individuals walk overground and on an instrumented treadmill. Gait Posture. 2021 Jan;83:174-176. doi: 10.1016/j.gaitpost.2020.10.025. Epub 2020 Oct 23. PMID 33152613
- [Background] Abbasi A, Yazdanbakhsh F, Tazji MK, Aghaie Ataabadi P, Svoboda Z, Nazarpour K, Vieira MF. A comparison of coordination and its variability in lower extremity segments during treadmill and overground running at different speeds. Gait Posture. 2020 Jun;79:139-144. doi: 10.1016/j.gaitpost.2020.04.022. Epub 2020 May 1. PMID 32408037
- [Result] Meyer A, Hrdlicka HC, Cutler E, Hellstrand J, Meise E, Rudolf K, Grevelding P, Nankin M. A Novel Body Weight-Supported Postural Perturbation Module for Gait and Balance Rehabilitation After Stroke: Preliminary Evaluation Study. JMIR Rehabil Assist Technol. 2022 Mar 1;9(1):e31504. doi: 10.2196/31504. PMID 35080495
- See also: Functional Gait Assessment. Shirley Ryan Ability Lab — https://www.sralab.org/rehabilitation-measures/functional-gait-assessment
- See also: Dynamic Gait Index. Shirley Ryan Ability Lab — https://www.sralab.org/rehabilitation-measures/dynamic-gait-index
- See also: Berg Balance Scale. Shirley Ryan Ability Lab — https://www.sralab.org/rehabilitation-measures/berg-balance-scale
- See also: Activities Specific Balance Confidence Scale. Shirley Ryan Ability Lab — https://www.sralab.org/rehabilitation-measures/activities-specific-balance-confidence-scale
- See also: Berg Balance Scale. Physio-pedia — https://www.physio-pedia.com/Berg_Balance_Scale

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred over 12 months, from October 2019 through September 2020. Participants were recruited from patients admitted to the inpatient stroke rehabilitation program at Gaylord Hospital after receiving a stroke diagnosis at a regional acute care hospital.
Pre-assignment Details: To be initially considered, patients had to be classified as a Moderate fall risk or better, shown by a Berg Balance Scale score of 21 or greater during their initial physical therapy evaluation. Patients who did not initially meet this criteria could screen-in at a later time pending a BBS reassessment. If the reassessment showed a sufficient functional improvement, and the patient had a discharge date of greater than two-weeks after the reassessment, the patient was recruited for the study.
Groups:
- Body Weight Support System Control Group: In this arm, participants will undergo their normal physical therapy treatment while using the ZeroG body weight support system.
  Body weight support system (BWSS) control group: The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
Period: Overall Study
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
Started | 16 | 16
Completed | 15 | 14
Not Completed | 1 | 2
Not completed — Early participant discharge from rehabilitation program after session 4 | 1 | 0
Not completed — Flare-up of existing orthopedic condition after session 4 | 0 | 1
Not completed — Acute ankle sprain after session 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Difference in numbers recruited versus analysed were due to the early discharge of 1 participant from the BWSS control group after session 4, the early withdrawal of 1 participant from the BWSS-P group after session 1 due to an acute ankle sprain, and the early withdrawal of 1 participant from the BWSS-P group after session 4 due to the flare-up of a preexisting orthopedic condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.38 (12.71) | 58.75 (15.43) | 58.56 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 13 | 12 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Difference in Berg Balance Scale Pre-intervention and Post-intervention Assessment Scores
Description: The Berg Balance Scale is a standardized objective measure of a subject/participant's balance. It is scored on a scale of 0 to 56, with 56 being the best score possible. Admission and discharge Berg scores are collected from a chart review within 48 hours of participant discharge. The change in Berg score is calculated by subtracting the participants admission or pre-assessment score from their discharge or post-assessment score: (Post assessment)-(Pre assessment)
Time Frame: The pre-assessment Berg Balance Scale score was collected during the initial physical therapy assessment within 48 hours of admission, as part of their normal care. The post-assessment was collected within 24 hours prior to discharge.
Population: The data from the 15 subjects from the BWSS control group and the 14 subjects from the BWSS-P who completed the study and were not withdrawn early, were included in this analysis.
Measure: Mean (Inter-Quartile Range); unit: Score on a Scale
Groups:
- Body Weight Support System Control Group (BBS Pre-score); Body Weight Support System Control Group (BBS Post-score): In this arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system. The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
- Body Weight Support System With Balance Perturbations (BBS Pre-score); Body Weight Support System With Balance Perturbations (BBS Post-score): Similar to the control group arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions. The BWSS with balance perturbations group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions. Additionally, this arm received eight balance perturbations, two in each direction (left lateral, right lateral, anterior, and posterior) each session. BWSS-P participants started at perturbation level "one" and progress up to level "ten" as appropriate. Each session, the perturbation level was set based on the participant's progress.
Arm/Group | Body Weight Support System Control Group (BBS Pre-score) | Body Weight Support System Control Group (BBS Post-score) | Body Weight Support System With Balance Perturbations (BBS Pre-score) | Body Weight Support System With Balance Perturbations (BBS Post-score)
Number analyzed (Participants) | 15 | 15 | 14 | 14
Score on a Scale | 30.20 [24 to 34] | 45.27 [40 to 53] | 30.43 [22.75 to 35.75] | 48.29 [43.50 to 53.50]
Statistical Analysis 1: Comparison: Body Weight Support System Control Group (BBS Pre-score) vs Body Weight Support System Control Group (BBS Post-score) vs Body Weight Support System With Balance Perturbations (BBS Pre-score) vs Body Weight Support System With Balance Perturbations (BBS Post-score); Null hypothesis for this analysis is that there will be no differences between pre-scores and post-scores across the different treatment arms. Prior to hypothesis testing, datasets were tested for normality using a Shapiro-Wilk test to inform if parametric or non-parametric testing was required; Test type: Superiority; p < 0.0001, Kruskal-Wallis — The a priori threshold for statistical significance was p<0.05. The p-value reported above was the calculated and resultant P-value for this analysis; Due sample size differences and pairwise nature of the data, a Kruskal-Wallis was conducted
Statistical Analysis 2: Comparison: Body Weight Support System Control Group (BBS Pre-score) vs Body Weight Support System Control Group (BBS Post-score); Null hypothesis for this comparison is that there would be no significant difference in the pre-score measurements between groups; Test type: Superiority; p = 0.0025, Dunn's Multiple Comparison Test — The a priori threshold for statistical significance was p<0.05. The p-value reported above was the calculated and resultant P-value for this analysis. The reported P-value is adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Body Weight Support System With Balance Perturbations (BBS Pre-score) vs Body Weight Support System With Balance Perturbations (BBS Post-score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0001, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Body Weight Support System Control Group (BBS Pre-score) vs Body Weight Support System With Balance Perturbations (BBS Pre-score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Body Weight Support System Control Group (BBS Post-score) vs Body Weight Support System With Balance Perturbations (BBS Post-score); Null hypothesis for this comparison would be that there would be no significant difference between post-scores of the two treatment groups; Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]

2. Primary Outcome: Comparison of Berg Balance Scale Assessment Score Changes
Description: The Berg Balance Scale is a standardized objective measure of a subject/participant's balance. It is scored on a scale of 0 to 56, with 56 being the best score possible. Admission and discharge Berg scores are collected using from a chart review within 48 hours of participant discharge. The change in Berg score is calculated by subtracting the participants admission or pre-assessment score from their discharge or post-assessment score: (Post assessment) - (Pre assessment). The score change between groups was then compared between the two treatment groups
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: Score on a Scale
Groups:
- Body Weight Support System Control Group: In this arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system. The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
- Body Weight Support System With Balance Perturbations: Similar to the control group arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions. The BWSS with balance perturbations group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions. Additionally, this arm received eight balance perturbations, two in each direction (left lateral, right lateral, anterior, and posterior) each session. BWSS-P participants started at perturbation level "one" and progress up to level "ten" as appropriate. Each session, the perturbation level was set based on the participant's progress.
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
Number analyzed (Participants) | 15 | 14
Score on a Scale | 15.07 [11.00 to 19.00] | 17.86 [9.00 to 24.50]
Statistical Analysis 1: Comparison: Body Weight Support System Control Group vs Body Weight Support System With Balance Perturbations; Null hypothesis is that there are no differences between groups. Prior to hypothesis testing, datasets were tested for normality using a Shapiro-Wilk test to inform if parametric or non-parametric testing was required; Test type: Superiority — Prior to analysis, the score change or difference between post-test and pre-test were calculated for each participant as: ScoreChange=(PostTest) - (PreTest). These changes in score were then compared; p = 0.3045, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Differences in the Percent Change of Berg Balance Scale (BBS) Assessment Scores
Description: The Berg Balance Scale is a standardized objective measure of a subject/participant's balance. It is scored on a scale of 0 to 56, with 56 being the best score possible. Admission and discharge Berg scores are collected using from a chart review within 48 hours of participant discharge. The BBS percent change is calculated using the following formula:
  [((Post assessement)-(Pre assessment))/(Pre assessment)] ×100%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: Percent Change
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
Number analyzed (Participants) | 15 | 14
Percent Change | 53.29 [29.27 to 66.67] | 66.95 [27.58 to 97.23]
Statistical Analysis 1: Comparison: Body Weight Support System Control Group vs Body Weight Support System With Balance Perturbations; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Prior to analysis, the score change or difference between post-test and pre-test were calculated for each participant as: PercentScoreChange = ([(PostTest)-(PreTest)]/[PreTest]) x 100%; p = 3152, Two-Tailed Welch t test — [p-value comment as in outcome 1, analysis 1]; Due to unequal standard deviation, a two-tailed Welch's t test was used

4. Primary Outcome: Activities-Specific Balance Confidence (ABC) Scale Score Change
Description: The ABC Scale subjectively measures a person's self-perceived balance-confidence to perform various tasks without losing balance or experiencing a sense of unsteadiness; it is based on a rating scale from 0% (no confidence) to 100% (completely confident); higher the score the better.
Time Frame: The pre-assessment ABC is completed at participant enrollment just prior to first intervention. The post-assessment ABC is completed immediately after final intervention.
Population: One participant in the Control group was discharged prior to completing the ABC post-assessment, resulting in an n=14.
Measure: Mean (Inter-Quartile Range); unit: Score on a Scale
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
Number analyzed (Participants) | 14 | 14
Score on a Scale | 20.57 [2.290 to 34.11] | 20.96 [6.793 to 35.16]
Statistical Analysis 1: Comparison: Body Weight Support System Control Group vs Body Weight Support System With Balance Perturbations; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9568, t-test, 2 sided — Prior to analysis, the score change between post assessment and pre-assessment was calculated. The threshold for significance was p<0.05; An unpaired T-test was used. Normality and F-test for Variances were conducted and found to be normal

5. Secondary Outcome: Toilet Transfer Score
Description: During their regular treatment, a modified functional independence measure, based on a scale of 0 (completely dependent) to 10 (completely independent), was used to assess each participant's assistance needs while undergoing toilet transfers. These scores were collected during a chart review conducted within 48 hours after participant discharge.
Time Frame: The pre-assessment Toilet transfer score is collected during the initial occupational therapy assessment within 48 hours of admission, as part of their normal care. The post-assessment is collected within 24 hours prior to discharge.
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: Score on a Scale
Groups:
- BWSS Control (Toilet Transfer Pre-Score); BWSS Control (Toilet Transfer Post-Score): In this arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system.
  The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
- BWSS-P (Toilet Transfer Pre-Score); BWSS-P (Toilet Transfer Post-Score): Similar to the control group arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions. The BWSS with balance perturbations group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions. Additionally, this arm received eight balance perturbations, two in each direction (left lateral, right lateral, anterior, and posterior) each session. BWSS-P participants started at perturbation level "one" and progress up to level "ten" as appropriate. Each session, the perturbation level was set based on the participant's progress.
Arm/Group | BWSS Control (Toilet Transfer Pre-Score) | BWSS Control (Toilet Transfer Post-Score) | BWSS-P (Toilet Transfer Pre-Score) | BWSS-P (Toilet Transfer Post-Score)
Number analyzed (Participants) | 15 | 15 | 14 | 14
Score on a Scale | 4.300 [4 to 4.5] | 7.7 [7 to 8] | 4.893 [4 to 5] | 8.393 [8 to 9]
Statistical Analysis 1: Comparison: BWSS Control (Toilet Transfer Pre-Score) vs BWSS Control (Toilet Transfer Post-Score) vs BWSS-P (Toilet Transfer Pre-Score) vs BWSS-P (Toilet Transfer Post-Score); Null Hypothesis, there would be no difference between the pre-score and post-score of each treatment group. Prior to hypothesis testing, datasets were tested for normality using a Shapiro-Wilk test to inform if parametric or non-parametric testing was required; Test type: Superiority; p < 0.0001, Kruskal-Wallis — [p-value comment as in outcome 1, analysis 1]; Due to the pairwise nature and abnormal distribution of the pre- and post-scores, a Kruskal Wallis test was completed
Statistical Analysis 2: Comparison: BWSS Control (Toilet Transfer Pre-Score) vs BWSS Control (Toilet Transfer Post-Score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: BWSS-P (Toilet Transfer Pre-Score) vs BWSS-P (Toilet Transfer Post-Score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: BWSS Control (Toilet Transfer Pre-Score) vs BWSS-P (Toilet Transfer Pre-Score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: BWSS Control (Toilet Transfer Post-Score) vs BWSS-P (Toilet Transfer Post-Score); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Ambulation Score
Description: During their regular treatment, a modified functional independence measure, based on a scale of 0 (completely dependent) to 10 (completely independent), was used to assess each participant's assistance needs while ambulating. These scores were collected during a chart review conducted within 48 hours after participant discharge.
Time Frame: The pre-assessment Ambulation score is collected during the initial occupational therapy assessment within 48 hours of admission, as part of their normal care. The post-assessment is collected within 24 hours prior to discharge.
Population: as for outcome 1
Measure: Mean (Full Range); unit: Units on a Scale
Groups:
- BWSS Control (Ambulation Pre-Score); BWSS Control (Ambulation Post-Score): In this arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system.
  The BWSS control group interventions consisted of various balance activities, including: marching, side-stepping, retro-ambulation, step-taps, and step-ups. The BWSS control group also practiced various gait tasks, including: ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.
- BWSS-P (Ambulation Pre-Score); BWSS-P (Ambulation Post-Score): Similar to the control group arm, participants underwent normal physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions. The BWSS with balance perturbations group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions. Additionally, this arm received eight balance perturbations, two in each direction (left lateral, right lateral, anterior, and posterior) each session. BWSS-P participants started at perturbation level "one" and progress up to level "ten" as appropriate. Each session, the perturbation level was set based on the participant's progress.
Arm/Group | BWSS Control (Ambulation Pre-Score) | BWSS Control (Ambulation Post-Score) | BWSS-P (Ambulation Pre-Score) | BWSS-P (Ambulation Post-Score)
Number analyzed (Participants) | 15 | 15 | 14 | 14
Units on a Scale | 4.357 [3 to 6] | 7.800 [6 to 9] | 4.750 [4 to 7] | 8.643 [6 to 10]
Statistical Analysis 1: Comparison: BWSS Control (Ambulation Pre-Score) vs BWSS Control (Ambulation Post-Score) vs BWSS-P (Ambulation Pre-Score) vs BWSS-P (Ambulation Post-Score); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Kruskal-Wallis — [p-value comment as in outcome 1, analysis 1]; Due to missing measurements and the pairwise nature of the pre- and post-scores, a Kruskal Wallis test was completed
Statistical Analysis 2: Comparison: BWSS Control (Ambulation Pre-Score) vs BWSS Control (Ambulation Post-Score); Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BWSS-P (Ambulation Pre-Score) vs BWSS-P (Ambulation Post-Score); Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BWSS Control (Ambulation Pre-Score) vs BWSS-P (Ambulation Pre-Score); Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BWSS Control (Ambulation Post-Score) vs BWSS-P (Ambulation Post-Score); Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Perturbation Level Progression
Description: All participants started at perturbation level "one" and progressed up to a maximum perturbation level of "ten" through the course of the study; the higher the level,the more intense the exerted force. The amount of force exerted at each perturbation level is pre-set by the manufacturer.The highest perturbation level achieved by the participant achieved was recorded immediately after each intervention session. In total, 8 readings were collected for each BWSS-P participant for the 8 intervention sessions completed for the study.
Time Frame: Perturbation level recordings completed for each of the 8 sessions completed over an average of 2 weeks.
Population: This outcome only includes observations from the BWSS-P group as the BWSS control did not receive perturbations. Values for each of the 8 study sessions are shown. The perturbation level for the 6th session for one subject was not recorded and was left blank.
Measure: Mean (Full Range); unit: Perturbation Level
Groups:
- BWSS-P (Perturbation Level Progression) Session 1; BWSS-P (Perturbation Level Progression) Session 2; BWSS-P (Perturbation Level Progression) Session 3; BWSS-P (Perturbation Level Progression) Session 4; BWSS-P (Perturbation Level Progression) Session 5; BWSS-P (Perturbation Level Progression) Session 6; BWSS-P (Perturbation Level Progression) Session 7; BWSS-P (Perturbation Level Progression) Session 8: As described in prior outcomes, BWSS-P participants underwent physical therapy treatment while using the ZeroG body weight support system, with the inclusion of 8 total balance perturbations each session, including 2 in the posterior, anterior, left lateral, and right lateral directions. BWSS-P group conducted the same balance and gait activities as the control group, including: marching, side-stepping, retro-ambulation, step-taps, step-ups, ambulation over the ground, going up and down stairs, and performing sit-to-stand transitions.In addition, this arm will receive eight balance perturbations, two in each direction (lateral, anterior, and posterior) each session. BWSS-P participants started at perturbation level "one" and progressed up to level "ten" as appropriate. Each session, the perturbation level was set based on the participant's progress. For this secondary outcome, the highest perturbation level achieved was recorded after each study session to track the progression of the BWSS-P participants.
Arm/Group | BWSS-P (Perturbation Level Progression) Session 1 | BWSS-P (Perturbation Level Progression) Session 2 | BWSS-P (Perturbation Level Progression) Session 3 | BWSS-P (Perturbation Level Progression) Session 4 | BWSS-P (Perturbation Level Progression) Session 5 | BWSS-P (Perturbation Level Progression) Session 6 | BWSS-P (Perturbation Level Progression) Session 7 | BWSS-P (Perturbation Level Progression) Session 8
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 14 | 14
Perturbation Level | 1.857 [1 to 4] | 3.143 [1 to 6] | 4.429 [2 to 7] | 4.929 [2 to 8] | 5.571 [3 to 10] | 6.077 [3 to 10] | 6.5 [4 to 10] | 6.875 [4 to 10]
Statistical Analysis 1: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 3 vs BWSS-P (Perturbation Level Progression) Session 4 vs BWSS-P (Perturbation Level Progression) Session 5 vs BWSS-P (Perturbation Level Progression) Session 6 vs BWSS-P (Perturbation Level Progression) Session 7 vs BWSS-P (Perturbation Level Progression) Session 8; Null hypothesis is there are no differences between groups. Prior to hypothesis testing, normality testing was conducted using a Shapiro-Wild test to inform if parametric or non-parametric testing was required; Test type: Superiority; p < 0.0001, Kruskal-Wallis — The threshold for statistical significance was p<0.05; Due to the missing measurement and the pairwise nature of the perturbation levels between participants, a Kruskal Wallis test was completed
Statistical Analysis 2: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 3 vs BWSS-P (Perturbation Level Progression) Session 4 vs BWSS-P (Perturbation Level Progression) Session 5 vs BWSS-P (Perturbation Level Progression) Session 6 vs BWSS-P (Perturbation Level Progression) Session 8; Null hypothesis for any comparisons would be that there is no significant mean perturbation level between sessions; Test type: Superiority; p > 0.9999, Dunn's Multiple Comparison Test — Reported p-value is adjusted for multiple comparisons. The a priori threshold for statistical significance was established as p<0.05; The p-value reported above was the result for 15 comparisons of the recorded perturbation levels in sessions: 1 vs 2, 2 vs 3, 3 vs 4, 3 vs 5, 3 vs 6, 4 vs 5, 4 vs 6, 4 vs 7, 4 vs 8, 5 vs 6, 5 vs 7, 5 vs 8, 6 vs 7, 6 vs 8, and 7 vs 8
Statistical Analysis 3: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 3; Test type: Superiority; p = 0.0629, Dunn's Multiple Comparison Test
Statistical Analysis 4: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 4; Test type: Superiority; p = 0.0069, Dunn's Multiple Comparison Test
Statistical Analysis 5: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 5; Test type: Superiority; p = 0.0003, Dunn's Multiple Comparison Test
Statistical Analysis 6: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 6; Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test
Statistical Analysis 7: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 7; Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test
Statistical Analysis 8: Comparison: BWSS-P (Perturbation Level Progression) Session 1 vs BWSS-P (Perturbation Level Progression) Session 8; Test type: Superiority; p < 0.0001, Dunn's Multiple Comparison Test
Statistical Analysis 9: Comparison: BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 4; Test type: Superiority; p = 0.6497, Dunn's Multiple Comparison Test
Statistical Analysis 10: Comparison: BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 5; Test type: Superiority; p = 0.0743, Dunn's Multiple Comparison Test
Statistical Analysis 11: Comparison: BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 6; Test type: Superiority; p = 0.0198, Dunn's Multiple Comparison Test
Statistical Analysis 12: Comparison: BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 7; Test type: Superiority; p = 0.0017, Dunn's Multiple Comparison Test
Statistical Analysis 13: Comparison: BWSS-P (Perturbation Level Progression) Session 2 vs BWSS-P (Perturbation Level Progression) Session 8; Test type: Superiority; p = 0.0006, Dunn's Multiple Comparison Test
Statistical Analysis 14: Comparison: BWSS-P (Perturbation Level Progression) Session 3 vs BWSS-P (Perturbation Level Progression) Session 7; Test type: Superiority; p = 0.5297, Dunn's Multiple Comparison Test
Statistical Analysis 15: Comparison: BWSS-P (Perturbation Level Progression) Session 3 vs BWSS-P (Perturbation Level Progression) Session 8; Test type: Superiority; p = 0.2595, Dunn's Multiple Comparison Test

8. Post Hoc Outcome: Sex Differences Between Treatment Arms
Description: The proportion of males and females between treatment arms was evaluated
Time Frame: This was conducted after the recruitment of the final participant.
Population: This analysis was completed using the information from the participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
Number analyzed (Participants) | 15 | 14
Participants
  Males | 13 | 10
  Female | 2 | 4
Statistical Analysis 1: Comparison: Body Weight Support System Control Group vs Body Weight Support System With Balance Perturbations; Null hypothesis was that there would be no difference in the proportion of males and females between treatment arms; Test type: Other — This is a descriptive analysis; p = 0.3898, Fisher Exact — Threshold for statistical significance was p<0.05; Odds Ratio (OR) = 2.600, 95% CI 2-sided [0.4671 to 15.300]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for the occurrence of adverse events over the course of the two-week period in which they were participating in the study. Due to the nature of the intervention, monitoring for adverse events after the treatment course was unnecessary.
Arm/Group | Body Weight Support System Control Group | Body Weight Support System With Balance Perturbations
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Body Weight Support System Control Group (N=16) | Body Weight Support System With Balance Perturbations (N=16)
Acute Ankle Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flare-up of pre-existing orthopedic condition (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was partly conducted during the early months of the COVID-19 pandemic (03/2020-08/2020). As such, this environment may have shortened the time participants were willing to spend in an inpatient setting. As a consequence, 40% of participants, at least once, needed to receive two sessions in the same day to complete all eight sessions due to expedited discharge timelines; in one case, a participant discharged before completing the last treatment session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT04919161/Prot_SAP_000.pdf